CLINICAL TRIAL: NCT02663128
Title: A Bioequivalence and Food Effect Study in Healthy Subjects Administered 2 Different Tablet Formulations of LY3314814
Brief Title: A Study of Lanabecestat (LY3314814) in Healthy Participants
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: AstraZeneca (Industry)
Collaborators: Eli Lilly and Company (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Basic Science
Other Study IDs: 16001; I8D-MC-AZEH (Other: Eli Lilly and Company)
Record Dates: First submitted 2016-01-21; First posted 2016-01-26 (Estimated); Results first posted 2019-03-22 (Actual); Last update posted 2019-11-01 (Actual); Status verified 2019-10

CONDITIONS: Healthy
MeSH Terms: interventions — lanabecestat

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (3):
- Lanabecestat Reference Fasted (Experimental): Lanabecestat: 50 mg administered once PO in each of 3 treatment periods.
  Interventions: Drug: Lanabecestat
- Lanabecestat Test Fasted (Experimental): Lanabecestat: 50 mg administered once PO in each of 3 treatment periods.
  Interventions: Drug: Lanabecestat
- Lanabecestat Test Non Fasted (Experimental): Lanabecestat: 50 mg administered once PO in each of 3 treatment periods.
  Interventions: Drug: Lanabecestat

INTERVENTIONS:
Drug: Lanabecestat — Administered orally
  Other Names: LY3314814; AZD3293

SUMMARY:
The purpose of this study is to measure how much of a new tablet formulation of lanabecestat gets into the blood stream and how long it takes the body to get rid of it, compared to the current tablet formulation of lanabecestat. The effect of a high fat meal on how quickly the body absorbs the new tablet formulation will also be evaluated. In addition any side effects of the study drug using both the new and current tablet formulations will be evaluated. The study will last about 22 days, with screening required within 30 days prior to the start of the study.

ELIGIBILITY:
Inclusion Criteria:

- Male participants: Will be sterile (including vasectomy) or agree to use an effective method of birth control and will not donate sperm during the study and for 3 months following the last dose of the investigational product

- Female participants: Women not of childbearing potential due to surgical sterilization or confirmed by medical history or menopause

- Are able to eat a high-fat, high-calorie meal within the defined time limit and abide by the food restrictions throughout the study

Exclusion Criteria:

* Have a history of or current, significant ophthalmic disease, as determined by the investigator or ophthalmologist
* Have vitiligo or any other clinically significant disorder of skin pigmentation as determined by the investigator or dermatologist
* History or presence of gastrointestinal, hepatic or renal disease or any other condition known to interfere with absorption, distribution, metabolism or excretion of drugs
* History of previous or ongoing psychiatric disease/condition
* Have an abnormality in the 12-lead electrocardiogram (ECG) that, in the opinion of the investigator, increases the risks associated with participating in the study, or have a history of significant dysrhythmias or atrioventricular (AV) block (including first degree AV block). Participants with history of persistent PR interval greater than (>)200 milliseconds (msec) will be excluded
* Have prolonged Fridericia-corrected QT interval (QTcF) of >470 msec
* Have a clinically significant abnormal blood pressure or heart rate (supine) as determined by the investigator
* Have a history of or current cardiovascular, respiratory, hepatic, renal, gastrointestinal, endocrine, hematological, or neurological disorders capable of significantly altering the absorption, metabolism, or elimination of drugs
* Are unwilling to comply with the dietary requirements/restrictions during the study
* Evidence of active renal disease (e.g, diabetic renal disease, polycystic kidney disease) or calculated creatinine clearance <50 milliliters per minute (mL/min)

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 18 (Actual)
Dates: Start 2016-01-31 (Actual); Primary Completion 2016-03-31 (Actual); Study Completion 2016-03-31 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Call 1-877-CTLILLY (1-877-285-4559) or 1-317-615-4559 Mon - Fri 9 AM - 5 PM Eastern time (UTC/GMT - 5 hours, EST), Study Director — Eli Lilly and Company

RESULTS

PARTICIPANT FLOW:
Recruitment Details: To obtain representative age-related data, attempts were made to enroll at least 6 participants who were >55 years of age.
Pre-assignment Details: Participants were randomized to 1 of 6 treatment sequences over 3 treatment periods that were 7 days long with a 7-day washout period between doses. Participants were either in a fasted state or fed state. Sequences contain a Reference (Fasted) dose; Test (Fasted) dose, and Test (Fed) dose: R (Fast)/ T (Fast)/ T (Fed), respectively.
Groups:
- Sequence 1: LY3314814 (AZD3293): 50 milligram (mg) administered once orally (PO) in each of 3 treatment periods. Treatment sequence: Reference (R [Fasted])/ Test (T [Fasted])/ T (Fed)
- Sequence 2: LY3314814 (AZD3293): 50 mg administered once PO in each of 3 treatment periods. Treatment sequence: T (Fasted)/T (Fed)/ R (Fasted)
- Sequence 3: LY3314814 (AZD3293): 50 mg administered once PO in each of 3 treatment periods. Treatment sequence:T (Fed)/ R (Fasted)/ T (Fasted)
- Sequence 4: LY3314814 (AZD3293): 50 mg administered once PO in each of 3 treatment periods. Treatment sequence:T(Fed)/ T (Fasted)/ R (Fasted)
- Sequence 5: LY3314814 (AZD3293): 50 mg administered once PO in each of 3 treatment periods. Treatment sequence: R (Fasted)/T (Fed)/ T (Fasted)
- Sequence 6: LY3314814 (AZD3293): 50 mg administered once PO in each of 3 treatment periods. Treatment sequence:T (Fasted)/ R (Fasted)/ T (Fed)
Period: Period 1
Arm/Group | Sequence 1 | Sequence 2 | Sequence 3 | Sequence 4 | Sequence 5 | Sequence 6
Started | 3 | 3 | 3 | 3 | 3 | 3
Received at Least One Dose of Study Drug | 3 | 3 | 3 | 3 | 3 | 3
Completed | 3 | 3 | 3 | 3 | 3 | 3
Not Completed | 0 | 0 | 0 | 0 | 0 | 0
Period: Period 2
Arm/Group | Sequence 1 | Sequence 2 | Sequence 3 | Sequence 4 | Sequence 5 | Sequence 6
Started | 3 | 3 | 3 | 3 | 3 | 3
Completed | 3 | 3 | 3 | 3 | 2 | 3
Not Completed | 0 | 0 | 0 | 0 | 1 | 0
Not completed — Physician Decision | 0 | 0 | 0 | 0 | 1 | 0
Period: Period 3
Arm/Group | Sequence 1 | Sequence 2 | Sequence 3 | Sequence 4 | Sequence 5 | Sequence 6
Started | 3 | 3 | 3 | 3 | 2 | 3
Completed | 3 | 3 | 3 | 3 | 2 | 3
Not Completed | 0 | 0 | 0 | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Population: Received at least one dose of study drug
Groups:
- 18 to 55 Years: LY3314814 (AZD3293): 50 mg administered once PO in each of 3 treatment periods. Reference formulation for fasted group Test formulation for fasted and non-fasted group
- > 55 Years: LY3314814 (AZD3293): 50 mg administered once orally PO in each of 3 treatment periods. Reference formulation for fasted group Test formulation for fasted and non-fasted group
- Total: Total of all reporting groups
Arm/Group | 18 to 55 Years | > 55 Years | Total
Number analyzed (Participants) | 8 | 10 | 18
Age, Continuous [Mean (Standard Deviation); unit: years] | 39.3 (9.9) | 61.4 (5.6) | 51.6 (13.6)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 1 | 4 | 5
  Male | 7 | 6 | 13
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 2 | 1 | 3
  Not Hispanic or Latino | 6 | 9 | 15
  Unknown or Not Reported | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 4 | 1 | 5
  White | 4 | 9 | 13
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 8 | 10 | 18

OUTCOME MEASURES:

1. Primary Outcome: Pharmacokinetics(PK): Maximum Concentration (Cmax) of LY3314814 (AZD3293)
Time Frame: Day 1 of Periods 1, 2, and 3: Predose, 0.5, 1, 1.5, 2, 3, 4, 6, 8, 12, 24, 36, 48, 56, 72, 96, and 120 hours post-dose
Population: All participants who received at least one dose of study drug and had evaluable PK data.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: nanogram per milliliter (ng/mL)
Groups:
- R (Fasted): LY3314814 (AZD3293): 50 mg administered once PO in each of 3 treatment periods. Reference formulation for fasted group
- T (Fasted): LY3314814 (AZD3293): 50 mg administered once PO in each of 3 treatment periods. Test formulation for fasted group.
- T (Fed): LY3314814 (AZD3293): 50 mg administered once PO in each of 3 treatment periods. Test formulation for non-fasted group
Arm/Group | R (Fasted) | T (Fasted) | T (Fed)
Number analyzed (Participants) | 18 | 17 | 18
nanogram per milliliter (ng/mL)
  18 to 55 Years | 194 (22) | 212 (22) | 164 (21)
  > 55 Years | 208 (31) | 196 (36) | 168 (32)

2. Primary Outcome: PK: Time of Maximum Observed Drug Concentration (Tmax) of LY3314814 (AZD3293)
Time Frame: Day 1 of Periods 1, 2, and 3:Predose, 0.5, 1, 1.5, 2, 3, 4, 6, 8, 12, 24, 36, 48, 56, 72, 96, and 120 hours post-dose
Population: All participants who received at least one dose of study drug and had evaluable PK data.
Measure: Median (Full Range); unit: Hour (h)
Arm/Group | R (Fasted) | T (Fasted) | T (Fed)
Number analyzed (Participants) | 18 | 17 | 18
Hour (h)
  18 to 55 Years | 2.00 [1.00 to 4.00] | 1.50 [1.00 to 3.02] | 4.01 [1.50 to 8.00]
  > 55 Years | 2.26 [1.00 to 4.12] | 1.50 [1.00 to 4.00] | 3.50 [1.50 to 6.00]

3. Primary Outcome: PK: Area Under the Concentration Versus Time Curve (AUC) of LY3314814 (AZD3293)
Time Frame: Day 1 of Periods 1, 2, and 3: Predose, 0.5, 1, 1.5, 2, 3, 4, 6, 8, 12, 24, 36, 48, 56, 72, 96, and 120 hours post-dose
Population: All participants who received at least one dose of study drug and had evaluable PK data.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: nanogram*hour/milliliter (ng*h/mL)
Arm/Group | R (Fasted) | T (Fasted) | T (Fed)
Number analyzed (Participants) | 18 | 17 | 18
nanogram*hour/milliliter (ng*h/mL)
  18 to 55 Years | 2920 (12) | 2850 (13) | 2970 (9)
  > 55 Years | 3040 (16) | 3020 (27) | 2820 (23)

ADVERSE EVENTS:
Description: Adverse events were analyzed and presented per respective formulation.
Arm/Group | R (Fasted) | T (Fasted) | T (Fed)
Serious Adverse Events (participants affected / at risk) | 0/18 | 0/17 | 0/18
Other Adverse Events (participants affected / at risk) | 5/18 | 4/17 | 4/18
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | R (Fasted) (N=18) | T (Fasted) (N=17) | T (Fed) (N=18)
Diarrhoea (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1)
Nausea (Gastrointestinal disorders) | 2 (2) | 0 (0) | 1 (1)
Upper respiratory tract infection (Infections and infestations) | 1 (1) | 0 (0) | 0 (0)
Arthralgia (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | 0 (0)
Back pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | 0 (0)
Pain in extremity (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | 0 (0)
Dizziness (Nervous system disorders) | 0 (0) | 2 (2) | 0 (0)
Headache (Nervous system disorders) | 1 (1) | 1 (3) | 3 (3)
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0)
Rhinorrhoea (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 0 (0)
Sneezing (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 0 (0)
Ecchymosis (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0) | 0 (0)
Pruritus (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of more than 60 days